CLINICAL TRIAL: NCT01079351
Title: A Sequential, Open-Label Study of the Pharmacokinetics and Safety of Intravenous Carbamazepine Relative to Oral Carbamazepine in Adult Patients With Epilepsy
Brief Title: A Study of the Pharmacokinetics (PK) and Safety of IV Carbamazepine Relative to Oral Carbamazepine in Adults With Epilepsy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lundbeck LLC (Industry)
Responsible Party: Lundbeck Inc., Lundbeck Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13103A; OV-1015 (Other: Former study ID)
Record Dates: First submitted 2010-03-01; First posted 2010-03-03 (Estimated); Last update posted 2010-04-23 (Estimated); Status verified 2010-04

CONDITIONS: Epilepsy
Keywords: Epilepsy; Intravenous Carbamazepine; Oral Carbamazepine
MeSH Terms: conditions — Epilepsy | interventions — Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Intravenous Carbamazepine — 10 mg/mL of intravenous Carbamazepine (CBZ) dissolved in 250 mg/mL of Captisol® (cyclodextrin) dosed at 70% of the patient's daily maintenance dose of oral CBZ administered after suitable dilution with D5W by intravenous infusion every 6 hours.
  Other Names: IV CBZ

SUMMARY:
The purpose of this study is to assess the safety, tolerability and steady-state pharmacokinetics of intravenous (IV) Carbamazepine (CBZ) infusions relative to orally administered CBZ in adult patients with epilepsy.

DETAILED DESCRIPTION:
This phase 1, multicenter, sequential, open-label study was designed to assess the safety, tolerability and pharmacokinetics of IV CBZ relative to orally administered CBZ in adult subjects with epilepsy. The study design used an increasing dose/treatment escalation cohort paradigm wherein subjects were enrolled in a cohort based on their total daily dose (TDD) of oral CBZ and their calculated creatinine clearance (CLcr; calculated by the Cockroft-Gault equation) on Day -28. The purpose of the increasing dose/treatment escalation cohort design was to provide a means for the independent data monitoring committee (IDMC) to assess safety prior to enrolling in subsequent cohorts; data were summarized by infusion time, renal function and dose. The initial subjects enrolled had normal renal function (CLcr >= 80 mL/min) and were stable on oral dosing of CBZ from 400 mg/day to 800 mg/day. Subsequent Dosing Cohorts enrolled subjects on higher doses of oral CBZ and allowed subjects with some renal impairment to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be diagnosed with any of the approved epilepsy indications for CBZ that include: Partial seizures with complex symptomatology (psychomotor, temporal lobe); Generalized tonic clonic seizures (grand mal); Mixed seizure patterns that include one of the above; Other partial or generalized seizures.
* Patient must be receiving a stable dose of oral CBZ (tablet or capsule formulation) for a minimum of 14 days prior to Day -28.
* Patient must be receiving a constant dose of all other concomitant medications / device (including AEDs, Vagal Nerve Stimulator (VNS), OTC medications, and herbal supplements) that may not interfere with the metabolism of CBZ for a minimum of 14 days prior to Day -28. No change in baseline AEDs are expected during the treatment period.
* The patient must be able to comply with maintaining an accurate epilepsy medication dosing diary and seizure diary.
* If female: Patient is not of childbearing potential.
* If childbearing potential: Must have a negative serum pregnancy test at Day -28 and a negative serum pregnancy test on Day -1; Must comply with a method of birth control acceptable to the investigator (with the exception of hormone based contraceptives which are contraindicated with the use of CBZ).

Exclusion Criteria:

* Patient is taking a daily oral dose of CBZ greater than 2000 mg per day.
* Patient is being treated with hormone based therapy for birth control.
* Patient has a QTc interval value that is greater than 450 msec.
* Patient has a screening ALT, AST or bilirubin > 3 times the upper limit of normal.
* Patients with CLCR < 30 mL/min or with a renal disorder (i.e. nephrotic syndrome, patients on hemodialysis or peritoneal dialysis or being considered for peritoneal or hemodialysis).
* Patient is receiving oral CBZ for absence seizures.
* Patient has had an episode of status epilepticus within 30 days of screening.
* Patient has a history of severe or serious adverse reactions to CBZ (e.g. aplastic anemia, agranulocytosis).
* Patient has been diagnosed with narrow angle glaucoma.
* Patient weighs less than 50 kg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2007-04; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To assess the safety, tolerability and pharmacokinetics of IV CBZ as a 30- and 15-minute infusion relative to orally administered CBZ in adult patients with epilepsy. | 31 days
To compare the steady-state pharmacokinetics of intravenously administered CBZ (Day 7) relative to orally administered CBZ (Day 0). | Day 7

SECONDARY OUTCOMES:
To assess the safety, tolerability and pharmacokinetics of IV CBZ when administered over a 2-5-minute infusion in a subset of patients. | 31 days
To assess the safety, tolerability and pharmacokinetics of IV CBZ in patients with mild or moderate renal impairment. | 31 days

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com

REFERENCES:
- [Derived] Lee D, Kalu U, Halford JJ, Biton V, Cloyd J, Klein P, Bekersky I, Peng G, Dheerendra S, Tolbert D. Intravenous carbamazepine as short-term replacement therapy for oral carbamazepine in adults with epilepsy: Pooled tolerability results from two open-label trials. Epilepsia. 2015 Jun;56(6):906-14. doi: 10.1111/epi.12991. Epub 2015 Apr 25. PMID 25912051